CLINICAL TRIAL: NCT00748033
Title: A Randomized, Single-blind, Cross-over, Single-centre Study in Healthy Volunteers Evaluating Subject Perception and Friction at Withdrawal of Catheters With Different Activation Times Compared to a Reference Catheter
Brief Title: A Study Evaluating a Urinary Catheter With Different Activation Times for the Wetting Solution, in Healthy Male Volunteers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wellspect HealthCare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: YA-CLO-0005
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Results first posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Urinary Catheterization

STUDY DESIGN:
Intervention Model Description: Two different activation times for the wetting solution for a urinary catheter will be used in healthy volunteers, compared to the use of a registered urinary catheter.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- LoFric POBE Hydro-Kit II, 5 seconds and then LoFric POBE Hydro-Kit II, 24 hours (Experimental): All subjects were first catheterizised with the reference catheter. After randomisation this group was first catheterizised with LoFric POBE Hydro-Kit II, activation time 5 seconds.
  Then the next test catheter was used LoFric POBE Hydro-Kit II, activation time 24 hours.
  Interventions: Device: Reference catheter: LoFric PVC, Nelaton 40 cm, CH 12; Device: LoFric POBE Hydro-Kit II, 5 seconds; Device: LoFric POBE Hydro-Kit II, 24 hours
- LoFric POBE Hydro-Kit II, 24 hours and then LoFric POBE Hydro-Kit II, 5 seconds (Experimental): All subjects were first catheterizised with the reference catheter. After randomisation this group was first catheterizised with LoFric POBE Hydro-Kit II, activation time 24 hours.
  Then the next test catheter was used LoFric POBE Hydro-Kit II, activation time 5 seconds.
  Interventions: Device: Reference catheter: LoFric PVC, Nelaton 40 cm, CH 12; Device: LoFric POBE Hydro-Kit II, 5 seconds; Device: LoFric POBE Hydro-Kit II, 24 hours

INTERVENTIONS:
Device: Reference catheter: LoFric PVC, Nelaton 40 cm, CH 12 — The subjects were first catheterized with this reference catheter.
Device: LoFric POBE Hydro-Kit II, 5 seconds — An unsalted LoFric POBE Hydro-Kit II, Nelaton 40 cm, CH 12 with sodium chloride in wetting solution, activation time 5 seconds
Device: LoFric POBE Hydro-Kit II, 24 hours — An unsalted LoFric POBE Hydro-Kit II, Nelaton 40 cm, CH 12 with sodium chloride in wetting solution, activation time 24 hours

SUMMARY:
The primary purpose of this study is to compare the subject's perception (separately for each randomized catheter) of practicing catheterization when using catheters with sodium chloride in wetting solution (using two different activation times) with a standard reference catheter. The hypothesis is that the subjects' perception of catheterization is the same or more positive when using the test catheters compared to the reference catheter.

DETAILED DESCRIPTION:
The study is designed as a randomized, single-blind, cross-over, single-centre, study in healthy male volunteers.

All subjects will first be catheterized with a reference catheter, which is proven to be well tolerated by most subjects. This catheter will be used as a reference catheter to be compared with the randomized catheters. One more reason for this first test is to withdraw subjects who cannot tolerate catheterizations. Subjects will qualify for the randomized part of the study only if the first catheterization could be performed without significant discomfort.

When the subject is randomized he will be catheterized with two urinary catheters in a randomized order during one day. The activation times for the wetting solution will be 5 seconds and 24 (± 2h) hours.

During each catheterization, the friction at withdrawal will be measured for the catheter using a Tension Test System.

The subjects will be blinded. 25 healthy volunteers will be recruited from a single centre in Sweden.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Healthy volunteer
* Male aged 18 years or over

Exclusion Criteria:

* Known or suspected, current impairment of and/or decreased urethral sensibility
* History of urethral morbidity
* History of urinary tract infection within three months, or ongoing symptomatic urinary tract infection
* Use of medications that may affect the urethra´s dryness (anti-cholinergic drugs or cortisone)
* Current drug, alcohol or other substance abuse
* Other significant disease or condition (e.g. benign prostate hypertrophy, other prostatic lesions), which may interfere with treatment and/or evaluation
* Allergy to antibiotics suspected poor compliance with the protocol during the complete study period

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Jacobsson, MD, PhD, Prof., Study Director — Dentsply Sirona Implants and Consumables
Locations (1):
- Karolinska Trial Alliance A2:01, Karolinska University Hospital, Stockholm, Sweden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a study with a crossover design between the test catheters. The subjects were first catheterized with a reference catheter and then catheterisized in a randomized order with the two test catheters.
  All subjects participated in all arms except one that participated only in 2 arms due to an adverse event.
  The subjects were catheterized three times during one day.. A minimum of two hours elapsed between the catheterizations and each catherization lasted for 3 minutes.
Groups:
- LoFric POBE Hydro-Kit II, 5 Seconds and Then LoFric POBE Hydro-Kit II, 24 Hours: Catheterizasion order:
  1. Reference Catheter, then washout for 2 hours
  2. LoFric POBE Hydro-Kit II activation time 5 seconds, then washout for 2 hours
  3. LoFric POBE Hydro-Kit II activation time 24 hours
- LoFric POBE Hydro-Kit II, 24 Hours and Then LoFric POBE Hydro-Kit II, 5 Seconds: Catheterizasion order:
  1. Reference Catheter, then washout for 2 hours
  2. LoFric POBE Hydro-Kit II activation time 24 hours, then washout for 2 hours
  3. LoFric POBE Hydro-Kit II activation time 5 seconds
Period: Overall Study
Arm/Group | LoFric POBE Hydro-Kit II, 5 Seconds and Then LoFric POBE Hydro-Kit II, 24 Hours | LoFric POBE Hydro-Kit II, 24 Hours and Then LoFric POBE Hydro-Kit II, 5 Seconds
Started | 12 | 13
Completed | 12 | 12 (One subject participated only in 2 arms due to an adverse event.)
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- LoFric POBE Hydro-Kit II, 5 Seconds and Then LoFric POBE Hydro-Kit II, 24 Hours: All subjects were first catheterizised with the reference catheter LoFric PVC, Nelaton 40 cm, CH 12.
  After randomisation this group was first catheterizised with LoFric POBE Hydro-Kit II, activation time 5 seconds.
  Then the next test catheter was used, LoFric POBE Hydro-Kit II, activation time 24 hours.
- LoFric POBE Hydro-Kit II, 24 Hours and Then LoFric POBE Hydro-Kit II, 5 Seconds: All subjects were first catheterizised with the reference catheter LoFric PVC, Nelaton 40 cm, CH 12.
  After randomisation this group was first catheterizised with LoFric POBE Hydro-Kit II, activation time 24 hours.
  Then the next test catheter was used LoFric POBE Hydro-Kit II, activation time 5 seconds.
- Total: Total of all reporting groups
Arm/Group | LoFric POBE Hydro-Kit II, 5 Seconds and Then LoFric POBE Hydro-Kit II, 24 Hours | LoFric POBE Hydro-Kit II, 24 Hours and Then LoFric POBE Hydro-Kit II, 5 Seconds | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 13 | 25
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.42 (6.10) | 26.17 (4.11) | 27 (5.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 13 | 25
Region of Enrollment [Number; unit: participants]
  Sweden | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Subjects' Perception at Insertion of Test Catheter Activated for 5 Seconds, Compared to Reference.
Description: The assessment was made in relation to the reference catheter, and the question to the subject was 'How do you experience this procedure/catheterization in comparison with the baseline procedure/catheterization regarding insertion?'.
Time Frame: A minimum of two hours elapsed between the catheterizations and each catherization lasted for 3 minutes. The subjects were catheterized three times during one day.
Population: The study was analysed using a per protocol approach only. One subject (Subject ID 125) was catheterized with the reference catheter and the catheter activated 24 hours, but not with the catheter activated 5 seconds. After discussions it has, however, been decided to use all available data. In conclusion all subjects fulfilling the inclusion criteria but none of the exclusion criteria were included in the Per-Protocol (PP) analysis set.
Measure: Number; unit: participants
Groups:
- LoFric POBE Hydro-Kit II, 5 Seconds: All subjects were first catheterizised with the reference catheter. After randomisation one group was first catheterizised with LoFric POBE Hydro-Kit II activation time 5 seconds, then the test catheter LoFric POBE Hydro-Kit II activation time 24 hours.
  The other group was first catheterizised with LoFric POBE Hydro-Kit II activation time 5 seconds, then test catheter LoFric POBE Hydro-Kit II activation time 24 hours.
Arm/Group | LoFric POBE Hydro-Kit II, 5 Seconds
Number analyzed (Participants) | 24
participants
  Very negative | 3
  Slightly negative | 10
  Same | 5
  Slightly positive | 6
  Very positive | 0
Statistical Analysis 1: Comparison: LoFric POBE Hydro-Kit II, 5 Seconds; Wilcoxon signed rank test, two-sided. Testing the hypothesis that the perception is same; Test type: Other; p = 0.0650, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Subjects' Perception at Insertion of Test Catheter Activated for 24 Hours, Compared to Reference.
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- LoFric POBE Hydro-Kit II, 24 Hours: All subjects were first catheterizised with the reference catheter then in a randomized order with the two test catheters.
Arm/Group | LoFric POBE Hydro-Kit II, 24 Hours
Number analyzed (Participants) | 25
Participants
  Very negative | 4
  Slightly negative | 8
  Same | 5
  Slightly positive | 7
  Very positive | 1
Statistical Analysis 1: Comparison: LoFric POBE Hydro-Kit II, 24 Hours; Wilcoxon signed rank test, two-sided. Testing the hypothesis that the perception is same; Test type: Other; p = 0.2487, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Subjects' Perception at Withdrawal of Test Catheter Activated for 5 Seconds, Compared to Reference.
Description: The assessment was made in relation to the reference catheter, and the question to the subject was 'How do you experience this procedure/catheterization in comparison with the baseline procedure/catheterization regarding withdrawal?'.
Time Frame: as for outcome 1
Population: Subjects fulfilling the inclusion criteria but none of the exclusion criteria were included in the Per-Protocol (PP) analysis set.
Measure: Count of Participants; unit: Participants
Groups:
- LoFric POBE Hydro-Kit II, 5 Seconds Hours: All subjects were first catheterizised with the reference catheter. After randomisation one group was first catheterizised with LoFric POBE Hydro-Kit II activation time 5 seconds, then the test catheter LoFric POBE Hydro-Kit II activation time 24 hours.
  The other group was first catheterizised with LoFric POBE Hydro-Kit II activation time 5 seconds, then test catheter LoFric POBE Hydro-Kit II activation time 24 hours.
Arm/Group | LoFric POBE Hydro-Kit II, 5 Seconds Hours
Number analyzed (Participants) | 24
Participants
  Very negative | 4
  Slightly negative | 6
  Same | 4
  Slightly positive | 8
  Very positive | 2
Statistical Analysis 1: Comparison: LoFric POBE Hydro-Kit II, 5 Seconds Hours; Wilcoxon signed rank test, two-sided. Testing the hypothesis that the perception is same; Test type: Other; p = 0.7288, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Subjects' Perception at Withdrawal of Test Catheter Activated for 24 Hours, Compared to Reference.
Description: as for outcome 3
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- LoFric POBE Hydro-Kit II, 24 Hours: All subjects were first catheterizised with the reference catheter. After randomisation one group was first catheterizised with LoFric POBE Hydro-Kit II activation time 5 seconds, then the test catheter LoFric POBE Hydro-Kit II activation time 24 hours.
  The other group was first catheterizised with LoFric POBE Hydro-Kit II activation time 5 seconds, then test catheter LoFric POBE Hydro-Kit II activation time 24 hours.
Arm/Group | LoFric POBE Hydro-Kit II, 24 Hours
Number analyzed (Participants) | 25
participants
  Very negative | 6
  Slightly negative | 6
  Same | 11
  Slightly positive | 2
  Very positive | 0
Statistical Analysis 1: Comparison: LoFric POBE Hydro-Kit II, 24 Hours; Wilcoxon signed rank test, two-sided. Testing the hypothesis that the perception is same; Test type: Other; p = 0.0045, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Comparison of the Perception at Insertion Between 5s and 24h Activation Times. Times
Description: Comparison of the perception at insertion between the catheters with 5s and 24h activation times.
Time Frame: as for outcome 1
Population: The study was analysed using a per protocol approach only.
Measure: Number; unit: participants
Groups:
- LoFric POBE Hydro-Kit II, 5 Seconds; LoFric POBE Hydro-Kit II, 24 Hours: All subjects were first catheterizised with the reference catheter LoFric PVC, Nelaton 40 cm, CH 12.
  After randomisation one group was first catheterizised with LoFric POBE Hydro-Kit II, activation time 5 seconds then LoFric POBE Hydro-Kit II, activation time 24 hours.
  After randomisation one group was first catheterizised with LoFric POBE Hydro-Kit II, activation time 2 hours then LoFric POBE Hydro-Kit II, activation time 5 seconds.
Arm/Group | LoFric POBE Hydro-Kit II, 5 Seconds | LoFric POBE Hydro-Kit II, 24 Hours
Number analyzed (Participants) | 24 | 24
participants
  Very negative | 3 | 3
  Slightly negative | 10 | 8
  Same | 5 | 5
  Slightly positive | 6 | 7
  Very positive | 0 | 1
Statistical Analysis 1: Comparison: LoFric POBE Hydro-Kit II, 5 Seconds vs LoFric POBE Hydro-Kit II, 24 Hours; Testing the hypothesis that 5s and 24 h are equal at insertion; Test type: Other; p = 0.4561, Wilcoxon (Mann-Whitney); Wilcoxon signed rank test if the difference between 5s and 24h is equal to 0

6. Secondary Outcome: Comparison of the Perception at Withdrawal Between 5s and 24h Activation Times.
Description: Comparison of the perception at withdrawal between the catheters with 5s and 24h activation times.
Time Frame: as for outcome 1
Population: The study was analysed using a per protocol approach only.
Measure: Number; unit: participants
Arm/Group | LoFric POBE Hydro-Kit II, 5 Seconds | LoFric POBE Hydro-Kit II, 24 Hours
Number analyzed (Participants) | 24 | 24
participants
  Very negative | 4 | 5
  Slightly negative | 6 | 6
  Same | 4 | 11
  Slightly positive | 8 | 2
  Very positive | 2 | 0
Statistical Analysis 1: Comparison: LoFric POBE Hydro-Kit II, 5 Seconds vs LoFric POBE Hydro-Kit II, 24 Hours; Testing the hypothesis that 5s and 24 h are equal at withdrawal; Test type: Other; p = 0.1797, Wilcoxon (Mann-Whitney); Wilcoxon signed rank test if the difference between 5s and 24h is equal to 0

7. Secondary Outcome: Test of Carry-over Effect at Insertion, Mean Rating of Perception on a Scale of 0 to 5
Description: The subjects perception of the catheterization will be classified as very negative, slightly negative, same, slightly positive or very positive.
  The mean perception of the 5s and the 24h catheter is calculated for each subject.
  The perception was measured on a scale from 1 (=very negative compared to the reference catheter) to 5 (=very positive compared to the reference catheter) and a 3 indicating that the perception was the same for the test catheter as for the reference catheter. Before doing any statistics all answers were reduced by 3 resulting in values from -2 (=very negative compared to the reference catheter) to +2 (=very positive compared to the reference catheter) and a 0 indicating that the perception was the same for the test catheter as for the reference catheter.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- 5s Followed by 24h; 24h Followed by 5s: Both groups were first catheterizied with the reference catheter. One group was then randomised to start with the catheter activated for 5 seconds followed by the catheter activated for 24 hours.
  The other group was randomised to start with the the catheter activated for 24 hours followed by the catheter activated for 5 seconds.
Arm/Group | 5s Followed by 24h | 24h Followed by 5s
Number analyzed (Participants) | 12 | 12
Scores on a scale | -0.17 (0.807) | -0.46 (0.865)
Statistical Analysis 1: Comparison: 5s Followed by 24h vs 24h Followed by 5s; The mean perception of the 5s and the 24h catheter is calculated for each patient. The patients are then divided in two groups depending on the order the patients received the two catheters and the hypotheses that the mean of the 5s and the 24h catheter is equal in the two groups are tested. If the test results in a significant p-value it can be concluded that a carry-over effect is present; Test type: Other; p = 0.5171, Wilcoxon (Mann-Whitney); Wilcoxon signed rank test if the difference between 5s and 24h is equal to 0

8. Secondary Outcome: Test of Carry-over Effect at Withdrawal, Mean Rating of Perception on a Scale of 0 to 5
Description: They had five alternative answers.The subjects perception of the catheterization will be classified as very negative, slightly negative, same, slightly positive or very positive.
  The mean perception of the 5s and the 24h catheter is calculated for each subject.
  The perception was measured on a scale from 1 (=very negative compared to the reference catheter) to 5 (=very positive compared to the reference catheter) and a 3 indicating that the perception was the same for the test catheter as for the reference catheter. Before doing any statistics all answers were reduced by 3 resulting in values from -2 (=very negative compared to the reference catheter) to +2 (=very positive compared to the reference catheter) and a 0 indicating that the perception was the same for the test catheter as for the reference catheter.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | 5s Followed by 24h | 24h Followed by 5s
Number analyzed (Participants) | 12 | 12
Score on a scale | -0.33 (0.835) | -0.33 (0.807)
Statistical Analysis 1: Comparison: 5s Followed by 24h vs 24h Followed by 5s; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.7105, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Tension Test System: Ref-24h Mean
Description: Tension test system (friction) at withdrawal. Comparison between the reference catheter and the 24 hours activation time. The MEAN for the withdrawal friction was measured in Newton (N).
Time Frame: The Tension test system was performed while withdrawing the catheters up to 5 seconds.
Population: The study was analysed using a per protocol approach only.
Measure: Mean (Standard Deviation); unit: Newton
Groups:
- MEAN Friction Value: Tension test system at withdrawal
Arm/Group | MEAN Friction Value
Number analyzed (Participants) | 24
Newton | 0.077 (0.088)
Statistical Analysis 1: Comparison: MEAN Friction Value; Test type: Other; p = 0.0003, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Tension Test System: Ref-24h Work
Description: Tension test system (friction) at withdrawal. Comparison between the reference catheter and the 24 hours activation time. The WORK for the withdrawal friction was measured in Joule (J).
Time Frame: The Tension test system was performed while withdrawing the catheters up to 5 seconds.
Population: The study was analysed using a per protocol approach only.
Measure: Mean (Standard Deviation); unit: Joule
Groups:
- Mean Friction Value: Mean Tension test system at withdrawal
Arm/Group | Mean Friction Value
Number analyzed (Participants) | 24
Joule | 0.011 (0.024)
Statistical Analysis 1: Comparison: Mean Friction Value; Test type: Other; p = 0.0346, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Tension Test System: Ref-5s MEAN
Description: Tension test system (friction) at withdrawal. Comparison between the reference catheter and the 5 seconds activation time. The MEAN for the withdrawal friction was measured in Newton (N).
Time Frame: The Tension test system was performed while withdrawing the catheters, up to 5 seconds.
Population: The study was analysed using a per protocol approach only.
Measure: Mean (Standard Deviation); unit: Newton
Arm/Group | MEAN Friction Value
Number analyzed (Participants) | 23
Newton | 0.073 (0.122)
Statistical Analysis 1: Comparison: MEAN Friction Value; Test type: Other; p = 0.0016, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Tension Test System: Ref-5s WORK
Description: Tension test system (friction) at withdrawal. Comparison between the reference catheter and the 5 seconds activation time. The WORK for the withdrawal friction was measured in Joule (J).
Time Frame: The Tension test system was performed while withdrawing the catheters, up to 5 seconds.
Population: The study was analysed using a per protocol approach only.
Measure: Mean (Standard Deviation); unit: Joule
Arm/Group | MEAN Friction Value
Number analyzed (Participants) | 23
Joule | 0.009 (0.030)

13. Secondary Outcome: Tension Test System: 24h-5s
Description: Tension test system (friction) at withdrawal. Comparison between the catheters with 24h activation time and the 5 seconds activation time.
  The MEAN for the withdrawal friction was measured in Newton (N).
Time Frame: The Tension test system was performed while withdrawing the catheters, up to 5 seconds.
Population: The study was analysed using a per protocol approach only.
Measure: Mean (Standard Deviation); unit: Newton
Arm/Group | MEAN Friction Value
Number analyzed (Participants) | 24
Newton | -0.013 (0.4092)

ADVERSE EVENTS:
Time Frame: Each subjects visited the clinic during one day. The subjects were catheterized for 3 minutes with each catheter. All subjects were catheterized with 3 catheters each, except one subject, who discontinued after test catheter 1 and was therefore only catheterized twice. At least 2 hours elapsed between each catheterization.
Description: In this study all adverse events will be judged as adverse device effect. Adverse events were not monitored during reference testing.
Arm/Group | LoFric POBE Hydro-Kit II, 5 Seconds | LoFric POBE Hydro-Kit II, 24 Hours
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 17/24 | 18/25
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LoFric POBE Hydro-Kit II, 5 Seconds (N=24) | LoFric POBE Hydro-Kit II, 24 Hours (N=25)
Discomfort during insertion of test catheter (Renal and urinary disorders) | 13 (13) | 12 (12)
Discomfort during withdrawal of test catheter (Renal and urinary disorders) | 10 (10) | 11 (11)
Discomfort during micturition after test catheter (Renal and urinary disorders) | 3 (3) | 2 (2)
Hematuria after test catheter is removed (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No